CLINICAL TRIAL: NCT02265328
Title: Efficacy of Combination Therapy of Glucocorticoids, and Bovine Colostrum in Treatment of Severe Alcoholic Hepatitis: A Pilot Study.
Brief Title: Efficacy of Combination Therapy of Glucocorticoids and Bovine Colostrum in Treatment of Severe Alcoholic Hepatitis.
Acronym: COBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dayanand Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Prof. Sandeep S Sidhu, Prof. Sandeep S sidhu, Dayanand Medical College and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COBS-2014
Record Dates: First submitted 2014-09-08; First posted 2014-10-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Severe Alcoholic Hepatitis in 'Extremis'- Defined by mDF>54
Keywords: Severe Alcoholic Hepatitis in 'Extremis'; Bovine Colostrum; Glucocorticoids
MeSH Terms: interventions — Enteral Nutrition; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bovine colostrum + prednisolone (Experimental): 1. Enteral nutrition: Protein 1.5 gm/kg/day, energy (kcal) 40/kg/day, carbohydrate 67-80%, Fat 20-33%.
  2. Oral prednisolone 40mg/day × 4 weeks and tapered to <40mg/day for next 4 weeks. If Lilli score > 0.45 after 7 days, then GC would be stopped and patients will be counselled for liver transplantation.
  3. Oral Bovine colostrum (200 ml (20 gram) TDS × 2 months.
  Interventions: Dietary Supplement: Bovine colostrum; Dietary Supplement: Enteral Nutrition; Other: prednisolone

INTERVENTIONS:
Dietary Supplement: Bovine colostrum — Oral Bovine colostrum 200 ml (20 gram) TDS × 2 months
Dietary Supplement: Enteral Nutrition — Enteral nutrition: Protein 1.5 gm/kg/day, energy (kcal) 40/kg/day, carbohydrate 67-80%, Fat 20-33%.
Other: prednisolone — Oral prednisolone 40mg/day × 4 weeks and tapered to <40mg/day for next 4 weeks. (If Lilli score > 0.45 after 7 days, then prednisolone would be stopped)
  Other Names: Wysolone, Predicort

SUMMARY:
Severe Alcoholic hepatitis (SAH), defined by modified Maddrey's Discriminant Function (DF) ≥32, is associated with significant morbidity and mortality. Of the various treatment modalities evaluated for treatment of SAH, corticosteroids have been the most extensively studied. Five out of 13 RCTs, and four out of 5 meta-analysis have shown a survival benefit with corticosteroids, especially in patients with DF ≥32 and/ or encephalopathy.However, the role of corticosteroids in SAH still remains somewhat controversial. Corticosteroid therapy is not considered the ideal option by all authors because their beneficial effect seems to be confined to a highly selected minority group in which the inhibitory effect of corticosteroids on liver inflammation is not outweighed by side effects such as weakened defence against infections, anti-anabolic effects, and possible ulcer promoting effects. Also corticosteroids are contraindicated in patients with renal failure, gastro-intestinal (GI) bleed, pancreatitis and active sepsis. Therefore, there have been constant efforts to evaluate new therapies for SAH. In a recent trial, combination of glucocorticoids plus N-acetylcysteine was found to improve one month survival in patients with SAH, compared with glucocorticoids alone. However the 6 month survival was not different in both groups.

Human Colostrum (HC) and Bovine Colostrum (BC) are rich in protein, immunoglobulin, lactoferrin and growth factors. Recent studies suggest that colostrum components, Lactroferrin, immunoglobulin and growth factor benefits physically active person and in treatment of autoimmune disorders. It is used for the treatment of a wide variety of gastrointestinal conditions, including non-steroidal anti-inflammatory drug-induced gut injury, H pylori infection, immune deficiency related diarrhea as well as infective diarrhea.

The guidelines by American College of Gastroenterology and other authors have suggested that a combination of CS and other drugs, which have different mechanisms of action, may be more beneficial for reducing mortality in SAH. Hence, we plan to conduct this pilot study to investigate the efficacy of a novel combination of corticosteroids, and Bovine colostrum in the treatment of SAH.

DETAILED DESCRIPTION:
Severe alcoholic hepatitis is associated with significant morbidity and mortality.

Diagnosis: The diagnosis of (AH) is made by the following criteria11

I.Chronic active alcohol abuse - > 80 grams in males and > 20 grams in females. II. Duration of jaundice < 3 months III. Serum Bilirubin >5 mg/dl IV. AST/ALT > 2:1 V. AST <500 IU/L, ALT <300 IU/L VI. Neutrophilic leucocytosis VII. Alcohol - non - alcohol index (ANI) determines the aetiology in an obese patient who drinks excessively. The ANI uses body mass index, mean corpuscular volume (MCV), AST/ALT ratio and gender to determine whether the aetiology is alcoholic steatohepatitis or non-alcoholic steatohepatitis (NASH). A high MCV, AST/ALT ratio > 1, low BMI and male gender favours alcohol as the aetiology, and this is reflected as a positive ANI score. A negative score implicates NASH as the cause of liver disease. The ANI calculator is available online (http://www.mayoclinic.org/girst/mayomodel10.html) VIII. Ethyl Glucuronide in urine12 detects alcohol intake within the last 3 days IX. Ethyl Glucuronide in hair13 detects intake of alcohol within the last few months X. Serum Enzyme linked immunosorbent Ethyl Glucuronide has a sensitivity and specificity of 92% and 91% respectively XI. Liver biopsy is useful when the diagnosis is uncertain and when corticosteroids are to be given for the treatment of SAH. A Transjugular liver biopsy is performed in most patients due to the coagulopathy in SAH.

Assessment of Severity Maddrey's Discriminant Function14 Discriminant Function Index (DFI) was originally described by Maddrey and colleagues in a placebo controlled study to assess the benefit of corticosteroids in patients with AH. The original formula was 4.6 x prothrombin time (PT) (seconds) + serum Bilirubin (mg/dl). It was observed that patients with a DFI >93 and treated with placebo had a 28 day survival of 25%, whereas those with a DFI < 93 had a 100% survival. Subsequently this score was modified in 19896 and called Modified Discriminant Function (MDF). MDF = 4.6 x (Patient's PT - Control PT) + serum bilirubin (mg/dl). Untreated patients with MDF >32 had a survival of 68%. The American College of Gastroenterology9 recommends that patients with MDF > 32 and / or Encephalopathy (SAH) be treated with Corticosteroids. The prothrombin time varies greatly depending on the sensitivity of the thromboplastin reagent used for the test. This is the drawback of the MDF.

MELD score15 The model for end stage liver disease (MELD) score predicts survival in patients with cirrhosis and is used to prioritize patients for liver transplantation.

MELD score = (0.957 x log serum creatinine + 0.378 x log serum bilirubin + 1.120 x log INR + 0.643) x 10. The advantage of MELD score is the use of INR in place of PT. The INR is comparable and uniform across laboratories worldwide. The American Association for Study of Liver Diseases (AASLD) recommends that a MELD score >20 predicts SAH and should be the criterion for initiating treatment. Serial monitoring of MELD score with a change of 2 or more points over the first week on treatment has independently predicted mortality.

GAHS score16 Glasgow Alcoholic Hepatitis Score (GAHS) includes age, peripheral Total Leucocyte Count, serum Bilirubin (at days 1 and 6-9), blood urea nitrogen and PT. It is a better predictor of mortality at 28 days than MDF. GAHS score > 9 has an extremely poor prognosis unless treated with Corticosteroids. The drawback is lack of international validation.

Child - Turcotte - Pugh score17 It is not traditionally used for predicting mortality of SAH. However, it helps to predict mortality at 3 and 6 months.

Treatment Abstinence from alcohol This is the most important factor in predicting the outcome after surviving the acute alcoholic hepatitis (AH) episode. The incidence of recidivism after recovery from the first episode of AH varies from 10 - 70 %.

Nutrition Enteral nutrition is the preferred mode for supplemental nutrition. It is cheap, maintains gut mucosal integrity. This in turn decreases the risk of bacterial and endotoxin translocation resulting in less infections and endotoxemia. Pooled data from 5 RCT's of AH have demonstrated improved nutritional status compared to standard dietary intake, but without improving survival rates.18 Pharmacotherapy Corticosteroids Corticosteroids (CS) are the most extensively used treatment for SAH. 6/13 RCT's and 4/6 meta-analysis have supported the use of CS in SAH. The last meta-analysis of individual patient data from 5 high quality RCT's using CS for SAH concluded that CS confers a 50% relative survival benefit at 1 month (85% versus 65% survival amongst those treated with CS versus untreated patients. The number of patients needed to treated (NNT) is 5 to reduce one death. Oral Prednisolone 40mg daily or parenteral methylprednisolone (for patients unable to take orally) 32 mg intravenously daily for 4 weeks is the standard therapy. The CS is tapered off over the next 4 weeks. A Lille score of >0.45 after 7 days of treatment with CS is an indication of non-response, increased susceptibility to infections and diminished survival19. The CS should be stopped if the lilli score is >0.45.

Pentoxifylline Pentoxifylline is a phosphodiesterase inhibitor. It is given orally in the dose of 400mg thrice a day for 28 days. In a pivotal study of 101 patients of SAH21, it was associated with survival benefit of 50%. In another study, it was found to be superior to CS20. In a recent study involving 50 patients at our center21, we found that 20% vs 40% mortality in patients treated with Pentoxifylline versus controls, after 4 weeks of treatment. Acute kidney injury was the cause of death in 20% compared to 70% patients in PTX group versus controls. PTX induces recovery of renal & hepatic functions with a trend towards increased survival. However, a metanalysis of 5 RCT failed to show any benefit with PTX22. The major adverse effects include vomiting, diarrhea, abdominal pain, headache and skin rash.

N-Acetylcyteine N-acetylcysteine could have value as an antioxidant in the treatment of acute alcoholic hepatitis, because the thiol group in N-acetylcysteine is able to reduce levels of free radicals. Administration of N-acetylcysteine might reconstitute the glutathione stocks of the hepatocytes.

At present, N-acetylcysteine is used in the treatment of acetaminophen induced hepatitis. Intravenous (I.V.) acetylcysteine is most often used as an antidote for acetaminophen overdose due to its ability to increase levels of glutathione; however, it is also used to treat non-acetaminophen-induced acute liver failure (NAI-ALF) and severe alcoholic hepatitis and to prevent contrast-induced nephropathy (CIN). Although the i.v. and oral formulations of acetylcysteine have been evaluated for these indications, most studies have examined the i.v. form. I.V. acetylcysteine is used in the treatment of NAI-ALF to improve oxygenation to the liver. A trial to evaluate the efficacy of glucocorticoids plus N-acetylcysteine, as compared with glucocorticoids alone, in patients with severe acute alcoholic hepatitis.23 reported improved one month survival in the combined treatment group. However the 6 month survival was not different in the two groups.

Bovine colostrum Human colostrum (HC) is the first milk produced after birth and is particularly rich in immunoglobulin (Ig), antimicrobial peptides (lactoferrin and lacto peroxidase) and other bioactive molecule, including growth factors which are important for nutrition, growth and development of newborn infants and also for passive immunity. Bovine colostrum (BC) is produced by the cows during the first 2 days post parturition. This "early" milk has nutrient profile and immunological composition substantially different from 'mature' milk. It contains macronutrient like proteins, carbohydrate, oligosaccharides, fats and micronutrients like vitamins and minerals, also growth factors, anti-microbial compounds and immune regulating constituents either not present in mature milk or present substantially in lower concentration.24,25 Historically colostrum has been used for various illnesses in India as well as abroad for thousands of years. Ayurvedic physicians of India have used bovine colostrum for both medicinal and spiritual purposes since cows were first domesticated. By the late 18th century, Western medicine started to take an interest in colostrum and study it for its potential health benefits. As a consequence, it was prescribed for many conditions, including immune system enhancement. Interestingly, until the development of penicillin and other artificial antibiotics in the 20th century, colostrum was commonly used for fighting bacterial infections. In the early 20th century it was noted that antibody levels in the first milk produced after birth were much higher than levels found in the milk that was produced 72 hours later. There are now over 2000 published scientific articles that document the safety and efficacy of using colostrum. This seemingly perfect food has been shown to be non-species specific26. In 2005, it was reported that is safe and effective in repair of tissues as well as for enhancing immunity.27 The use of bovine colostrum as dietary supplement has increased substantially over the past decades. Bovine colostrum is harvested within first few hours of calving from dairy animals. The herds of cows are kept under close supervision in good state of hygiene without exposure to antibodies, pesticides and anithelmintic. They are monitored according to FDA criteria. The colostrum collected within 24 hours contains maximum substances but less in amounts, colostrum collected later will be more but contain less immunoglobins.27 Colostrum contains the growth factors that help build lean muscle, including insulin-like growth factors (IGF-I & IGF-II) and growth hormone (GH). IGF-I, which is found naturally in colostrum, is the only natural hormone capable of promoting muscle growth by itself. The IGFs in humans and cows are identical, but bovine colostrum actually contains a greater concentration of IGF-I than human colostrum. This fact makes bovine colostrum attractive to bodybuilders, athletes and others seeking to gain muscle mass. According to a study conducted in Finland, IGF-1 induces protein synthesis, which leads to an increase in lean muscle mass without a corresponding rise in adipose (fat) tissue. The growth factors in colostrum "shift fuel utilization from carbohydrate to fat. It mean that body will burn more fat, including fat made from the carbohydrate and protein that are consumed, producing fuel more efficiently.28 Bovine has hormone factor like gastrin which plays a role as a trophic factor for mucosal growth with in stomach. GLP-2 has shown a general trophic response with in the gut.

Peptide growth factors in colostrum can influence the maintenance of mucosal mass and integrity. EGF stimulates cell proinfection and also influences crypt fission.

Human colostrum has higher concentration of growth factors as compared to bovine colostrum. The tables and figure below indicate how HC and BC differ in their nutrient content, immunological factors and growth factors (Table 1, 2,3)

While BC are considered a rich source of Ig, growth factors, and lactoferrin, currently no specific standards exist that define BC dietary supplements with respect to actual constituents or amounts of constituents. The following constituents are generally present in bovine colostrums: macronutrients; vitamins; minerals; Ig (IgG, IgM, and IgA - including the secretory form); cytokines including interleukin-1beta (IL-1β), interleukin- 6 (IL-6), tumor necrosis factor-alpha (TNF-α), and interferon-gamma (INF-γ); growth factors including insulin-like growth factor (IGF) I and II, transforming growth factor-beta (TGF-β), and epidermal growth factor; lactoperoxidase; and lactoferrin. Depending on the health of the cows, feeding practices followed, collection period, and the processing/concentration practices utilized by specific manufacturers, the actual range and quantities of specific macro- and micronutrients, Ig, cytokines, growth factors, and other compounds might vary considerably.

BC contain relatively high amounts of Ig. Typically, Ig in general, and IgG specifically, constitutes the largest contribution to protein content in BC, with lactalbumin and casein contributing lesser amounts. Mean percentages of fat, protein, and lactose in colostrum were 6.7, 14.9, and 2.5, respectively. Other reports have estimated Ig concentrations from bovine mammary secretions with ranges for IgG1 (52-87 g/L), IgG2 (1.6-2.1 g/L), IgM (3.7-6.1 g/L), and IgA (3.2-6.2 g/L).35 As a rule, the Ig contribution will decline substantially in any BC collected more than 24 hours post-parturition and the amount of lactalbumin and casein will increase proportionately.

Table : Immunoglobulin Composition during the first 10 hours post parturition

Constituents Concentration (g/L) IgG 30.4 IgA 3.5 IgM 9.6

Detailed research plan (Materials and Methods) Study design and setting Twenty five Patients will be enrolled in this pilot study. The study will be conducted on patients of Severe Alcoholic Hepatitis admitted in the Department of Gastroenterology, Dayanand Medical College and Hospital, Ludhiana. Informed consent shall be taken from the patient/nearest relative of the patient for enrollment in the trial.

Study population

Inclusion Criteria:

1. Severe Alcoholic hepatitis (mDF > 32) 2. Age 18-65 Years 3. DF>32 4. Actively consuming alcohol within 6 weeks of entry into the study Exclusion Criteria

1. Failure to obtain informed consent
2. Active infection or sepsis
3. Other concomitant causes of liver disease: viral hepatitis, autoimmune liver disease, metabolic liver disease, vascular liver disease
4. HIV positive
5. Cow milk allergy or severe lactose intolerance
6. Active Gastrointestinal bleeding
7. Acute kidney injury at time of randomization with Creatinine > 1.5 mg/dL
8. Evidence of acute pancreatitis or biliary obstruction
9. Subjects who are pregnant or lactating
10. Significant systemic cardio-pulmonary illness
11. Patients requiring the use of vasopressors or inotropic support in 12 hours prior to randomization
12. Treatment for alcoholic hepatitis within 1 month of study entry with corticosteroids use>1 week.
13. Any patient who has received any investigational drug or device within 30 days entering into the study.

Study Methods Enrolment of patients, assessing eligibility and obtaining informed consent will be carried out by one of the investigators (S.S. Sidhu, O. Goyal) Study Intervention

Treatment for SAH:

1. Enteral nutrition: Protein 1.0-1.5 gm/kg/day, energy (kcal) 30-40/kg/day, carbohydrate 67-80%, Fat 20-33%.
2. Steroids were administered according to protocol. The initial dose of methyl prednisolone (40 mg/day) for one month was tapered to (<40 mg/day) for one month.

   If Lilli score > 0.45 after 7 days, then GC would be stopped and patients will be counselled for liver transplantation.
3. Oral BC (200 ml (20 gram/day) TDS × 8 weeks.

Laboratory tests Biochemical tests Hemogram, blood glucose, liver function tests, prothrombin time, serum electrolytes, blood urea and serum creatinine will be done at baseline, and at 2nd and 7th day of treatment, or earlier if indicated. AFP and Lipase will be done at admission.

Microbiologic tests:

A diagnostic paracentesis will be done in all patients with ascites, at baseline, to diagnose Spontaneous Bacterial Peritonitis. A repeat cell count (Total and differential) shall be done on day 7 in patients diagnosed to have Spontaneous Bacterial Peritonitis. Blood culture, urine culture, cultures of aspirates from endotracheal tubes in ventilated patients for aerobic and anerobic bacteria, and fungi shall be done on at admission. A chest radiograph shall also be done.

Tests for etiologic evaluation:

Etiology of cirrhosis will be taken as alcohol if there is a history of significant alcohol intake (20-40 gm/day for females, and 60-80 gm/day for males for 10 years or more). Each patient will be tested for Hepatitis B surface antigen (HbsAg) and Anti-hepatitis C (HCV) antibody using a third generation commercial ELISA. Wherever indicated, autoimmune hepatitis will be diagnosed using antinuclear antibody, anti-smooth muscle antibody and anti-LKM; and hemochromatosis using serum iron, TIBC, ferritin and transferrin saturation. Each patient shall have an abdominal ultrasonography. Upper gastrointestinal endoscopy would be done, if indicated.

Outcome measures and endpoints

Primary outcome measure

(a) Change in mDf at 2 month

Secondary outcome measures

1. Survival at 1 month
2. Survival at 2 month

Study Endpoints

1. Liver related death
2. Death due to other causes
3. Discontinuation due to adverse effects
4. Discharge from hospital

Monitoring for Adverse Events:

Any adverse event will be recorded specifying the time of onset, the duration, the severity and the relationship to the test medication.

Tolerability Tolerability of the study drug will be assessed by comparison of full blood cell count, liver function tests and renal function tests at baseline and at end of treatment.

Follow-up All patients will be followed up until recovery.

Statistical Analysis:

Data will be present as means+ SD for quantitative variables and percentage for qualitative variables. The change in the mDf score and Lille score with in the group will be assessed by analysis of variance. A P- value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Severe Alcoholic hepatitis (mDF > 54)
2. Age 18-65 Year

4. Actively consuming alcohol within 6 weeks of entry into the study

Exclusion Criteria:

1. Failure to obtain informed consent
2. Active infection or sepsis
3. Other concomitant causes of liver disease: viral hepatitis, autoimmune liver disease, metabolic liver disease, vascular liver disease
4. HIV positive
5. Cow milk allergy or severe lactose intolerance
6. Active Gastrointestinal bleeding
7. Acute kidney injury at time of randomization with Creatinine > 1.5 mg/dL
8. Evidence of acute pancreatitis or biliary obstruction
9. Subjects who are pregnant or lactating
10. Significant systemic cardio-pulmonary illness
11. Patients requiring the use of vasopressors or inotropic support in 12 hours prior to randomization
12. Treatment for alcoholic hepatitis within 1 month of study entry with corticosteroids use>1 week.
13. Any patient who has received any investigational drug or device within 30 days entering into the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in mDf Value from baseline to 8 weeks | 2 month

SECONDARY OUTCOMES:
Change in Endotoxin level from baseline to 8 weeks | 2 month
Cytokines Levels (αTNF, IL 6, IL 8) from baseline to 8 weeks. | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep S Sidhu, MD,DM, Principal Investigator — Dayanand Medical College and Hospital; Omesh Goyal, MD,DM, Principal Investigator — Dayanand Medical College and Hospital
Locations (1):
- Dyanand Medical College and Hospital, Ludhiana, Punjab, India